CLINICAL TRIAL: NCT06391385
Title: The Effects of Temporary Ileostomy on Outcome in Patients With Rectal Cancer, A Prospective Comparative Cohort Study
Brief Title: The Effects of Temporary Ileostomy on Outcome in Patients With Rectal Cancer
Acronym: Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tishreen_ Temporary Ileostomy
Record Dates: First submitted 2024-01-04; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: Rectal cancer; ileostomy; morbidity; anterior rectal resection
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The surgical procedure was performed by laparotomy, with resection of the rectum and mesorectum (TME) up to the level of the pelvic diaphragm, sparing the autonomic nerves. End-to-end anastomosis was performed either with a stapler or by hand-sewn. Patients were assigned to group I (19 patients) who had undergone temporary ileostomy, and group II (28 patients) who didn't undergo ileostomy. Patients were followed up at regular intervals and outcomes were compared between two groups.
Masking Description: No blinding or masking is implemented in this open-label study. Both participants and healthcare providers are aware of the intervention status. This design allows for transparency in the treatment approach, and outcomes will be assessed without blinding. The lack of masking is a characteristic of the study design and does not impact the validity of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Ileostomy Arm (No Intervention): Participants in this arm do not undergo the intervention of a protective ileostomy. The management for this group involves. The outcomes for this arm will be assessed in comparison to the group that receives the protective ileostomy. This arm serves as the control/comparative group to evaluate the impact of the intervention on the specified outcomes.
- Ileostomy Arm (Experimental): Ileostomy Arm Description: Participants in this arm undergo the intervention of a protective ileostomy. The surgical procedure involves. This arm serves as the experimental group to evaluate the impact of the protective ileostomy on specified outcomes. The outcomes for this arm will be compared to those in the non-interventional (comparative) arm to assess the effectiveness and potential benefits of the ileostomy intervention.
  Interventions: Procedure: protective ileostomy

INTERVENTIONS:
Procedure: protective ileostomy — Preparation of the bowel was performed before surgery with the administration of intravenous perioperative antibiotic prophylaxis. The surgical procedure was performed by laparotomy, with resection of the rectum and mesorectum (TME) up to the level of the pelvic diaphragm, sparing the autonomic nerves. End-to-end anastomosis was performed either with a stapler or by hand-sewn.
  Arms: Ileostomy Arm

SUMMARY:
The purpose of this prospective comparative cohort study was to assess the effect of protective ileostomy on the outcomes of patients with rectal cancer who underwent low anterior rectal (LAR) resection in patients with a diagnosis of colorectal cancer of both sexes and all ages that required low anterior resection(LAR) attending the Department of General Surgery at Tishreen University Hospital in Lattakia-Syria during the two years (May 2021- May 2023). the main question to answer is does protective ileostomy reduce leakage, SSI rate, and duration of hospitalization in patients with colorectal cancer. . Patients are divided into two groups: group 1: patients who underwent ileostomy (19 patients), and group 2 is the comparative group: patients who didn't (28 patients). Morbidity and mortality were compared between the two groups, to study the outcomes of protective ileostomy

DETAILED DESCRIPTION:
Anastomotic leakage is encountered frequently after colorectal cancer (CRC) surgery, which is considered one of the potentially lethal complications, affecting the quality of life and increasing hospital costs. The role of a protective stoma has been debated. Therefore, The purpose of this study was to assess the effect of protective ileostomy on the outcomes of patients with rectal cancer who underwent low anterior rectal (LAR) resection.

This is a prospective comparative study of a group of patients with a diagnosis of colorectal cancer of both sexes and all ages that required low anterior resection(LAR) attending the Department of General Surgery at Tishreen University Hospital in Lattakia-Syria during the two years (May 2021- May 2023). The exclusion criteria were patients who underwent abdominoperineal resection with permanent ileostomy. The following workup included: a history and physical examination.

Preparation of the bowel was performed before surgery with the administration of intravenous perioperative antibiotic prophylaxis. The surgical procedure was performed by laparotomy, with resection of the rectum and mesorectum (TME) up to the level of the pelvic diaphragm, sparing the autonomic nerves. End-to-end anastomosis was performed either with a stapler or by hand-sewn. Patients were assigned to group I (19 patients) who had undergone temporary ileostomy, and group II (28 patients) who didn't undergo ileostomy. Patients were followed up at regular intervals and outcomes were compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of colorectal cancer that required low anterior resection(LAR)
* Both sexes
* All ages
* Attending the Department of General Surgery at Tishreen University Hospital in Lattakia-Syria during the two years (May 2021- May 2023).

Exclusion Criteria:

* Patients who underwent abdominoperineal resection with permanent ileostomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The Rate of Anastomosis leakage | up to 2 weeks post operatively
  Anastomosis leakage is defined as the unintended escape of gastrointestinal contents from the site of surgical anastomosis, typically occurring after a low anterior rectal (LAR) resection. It is a critical postoperative complication that can lead to various adverse effects, including peritonitis, abscess formation, and increased morbidity. The evaluation of anastomosis leakage involves careful monitoring for clinical signs, diagnostic imaging, and, if necessary, interventions such as reoperation or drainage procedures. The occurrence and management of anastomosis leakage serve as a key primary outcome measure in this study, contributing valuable insights into the efficacy and safety of the protective ileostomy intervention
The Rate of Surgical Site Infection | up to 6 weeks post operatively
  Surgical Site Infection is a postoperative complication characterized by the invasion of microorganisms into the surgical incision or the deeper tissues surrounding the operative site. In the context of this study, the evaluation of SSI involves monitoring for clinical signs of infection, such as redness, swelling, warmth, or discharge, and may require additional diagnostic assessments. The occurrence of Surgical Site Infection is a critical parameter, impacting patient recovery, healthcare costs, and overall postoperative morbidity. As a primary outcome measure, the study aims to comprehensively assess the incidence and characteristics of SSI, providing crucial insights into the effectiveness of the protective ileostomy intervention.

OTHER OUTCOMES:
The Duration of surgery | from open incision to skin until closing the skin during the operaton
  The Duration of Surgery is a critical parameter measured from the initiation of the surgical incision to the closure of the incision. This outcome is pivotal in understanding the efficiency and complexity of the surgical procedure. It encompasses the time required for key stages, such as tumor resection, anastomosis, and closure. A shorter duration may indicate a more streamlined and less invasive procedure, potentially contributing to reduced patient morbidity and improved postoperative outcomes. Monitoring the Duration of Surgery as a primary outcome provides valuable insights into the procedural intricacies and overall efficiency of the interventions, aiding in the evaluation of the protective ileostomy's impact on surgical timelines.
The Duration of Hospitalization | from day 0 post surgery until discharge from the hospital , up to 4 weeks
  The Duration of Hospitalization refers to the total time a patient spends in the hospital after undergoing low anterior rectal (LAR) resection with or without protective ileostomy. This outcome is crucial in assessing the postoperative recovery period and resource utilization. A shorter duration may indicate a smoother recovery and reduced postoperative complications, potentially contributing to decreased healthcare costs. Monitoring the Duration of Hospitalization as a primary outcome provides essential information about the impact of protective ileostomy on the length of hospital stay, aiding in the evaluation of its influence on patient recovery and healthcare resource management.

CONTACTS AND LOCATIONS:
Locations (1):
- Tishreen University, Latakia, Syria

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT06391385/Prot_SAP_000.pdf